CLINICAL TRIAL: NCT01091077
Title: A Pilot Study of the Grapefruit Flavonoid Naringenin for the Treatment of HCV Infection
Brief Title: A Pilot Study of the Grapefruit Flavonoid Naringenin for HCV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Harvard University (Other)
Responsible Party: Principal Investigator, Arthur Y. Kim, MD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GFN-001
Record Dates: First submitted 2010-03-17; First posted 2010-03-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C Virus; HCV Infection; Chronic HCV; Hepatitis C
Keywords: dietary supplement
MeSH Terms: conditions — Hepatitis C | interventions — naringenin; grapefruit seed extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Naringenin (Placebo Comparator): Single dose of naringenin, compared to placebo in the same individual.
  Interventions: Dietary Supplement: Naringenin

INTERVENTIONS:
Dietary Supplement: Naringenin — 1 gram of naringenin mixed with 16 grams of hydroxypropyl-β-cyclodextrin in 250 mL of water
  Other Names: Grapefruit

SUMMARY:
Hepatitis C virus when it leaves the cells in the liver is bound to a type of fat. An component of grapefruit could block this fat and thus lower the amount of virus in the blood stream. We propose that treatment with this ingredient, called naringenin, could be used to block this fat and HCV in persons infected with hepatitis C.

DETAILED DESCRIPTION:
The hepatitis C virus is actively secreted by the liver of infected patients while bound to very low density lipoprotein (vLDL). The grapefruit flavonoid naringenin could be used to block vLDL secretion and lower the circulating viral titer.

Hypothesis:

Treatment with naringenin will block vLDL and HCV secretion in persons infected with HCV.

Primary Objective

To study the safety and pharmacokinetics of a single-dose of naringenin

Secondary Objectives

1. To study the changes in circulating HCV titers during the transition from a fasted to fed state.
2. To study the changes in circulating HCV titers after administration of the grapefruit flavonoid naringenin.
3. To study effects of naringenin on vLDL secretion.

This is a single-arm, cross over study where placebo is administered during a transition from a fasted to a fed state, then the protocol is repeated with a single dose of naringenin plus cyclodextrin, using the previous measurements as his/her own control

ELIGIBILITY:
Inclusion Criteria:

* HCV infection as documented by any licensed ELISA test kit any time prior to study entry.
* Documentation of chronic high-titer HCV infection, as defined as a positive HCV viral load >400,000 IU/ML measured within 2 years prior to study entry and after the last interferon-based treatment course.
* HCV genotype - all genotypes are eligible for this trial
* Prior (but not current) treatment with interferon-based therapies are allowed
* Subjects with documented or suspected hepatic cirrhosis must have a Modified Child-Pugh-Turcotte (CPT) Score of 5 or less within 42 days prior to study entry.

Exclusion Criteria:

* Presence of known causes of significant liver disease including chronic or acute hepatitis B, acute hepatitis A, autoimmune hepatitis, hemochromatosis, or homozygote alpha-1 antitrypsin deficiency.
* Evidence of decompensated liver disease manifested by presence of or history of ascites, variceal bleeding, or hepatic encephalopathy, and/or a Child-Pugh score of 6 or higher.
* History of major organ transplantation, including liver, with an active, functioning graft
* Candidates for liver transplant, as evidenced by active listing
* Receipt of HCV treatment within 28 days prior to study entry.
* Breast-feeding.
* Pregnancy, or considering getting pregnant within 1 month
* Use of lipid-lowering drugs (i.e. HMG-CoA reductase inhibitors, fibrates, omega-3 fatty acids, bile acid sequestrants, ezetimibe, and niacin derivatives), within 3 months prior to study entry
* Use of drugs with known interactions with grapefruit juice
* Known HIV infection
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* History of an adverse reaction to citrus fruits
* History of uncontrolled seizure disorder.
* Uncontrolled depression or other psychiatric disorder such as untreated Grade 3 psychiatric disorder, Grade 3 disorder not amenable to medical intervention, or any hospitalization within the past 52 weeks that in the opinion of the site investigator might preclude tolerability of study requirements.
* History of autoimmune processes, including but not limited to Crohn's disease, ulcerative colitis, severe psoriasis, rheumatoid arthritis, that have been exacerbated by previous interferon use.
* Any systemic antineoplastic or immunomodulatory treatment or radiation within 24 weeks prior to study entry.
* Serious illness including malignancy, active symptomatic coronary artery disease within 24 weeks prior to study entry, or other chronic medical conditions that may preclude completion of the protocol in the investigator's opinion.
* Past history of estrogen-responsive breast cancer
* Use of antidiabetic medications within 12 weeks prior to study entry.
* Fasting plasma glucose ≥126 mg/dL within 42 days prior to study entry or currently or previously treated at any time for diabetes with measures other than diet. NOTE: Women with a history of gestational diabetes not requiring any treatment for diabetes before or after pregnancy are eligible for participation. Subjects with diabetes/hyperglycemia occurring in the context of short-term use of corticosteroids, growth hormone, or other diabetogenic medication, but not requiring any treatment for diabetes after discontinuation of the implicated medication, are eligible to participate. Subjects with diabetes/hyperglycemia following an episode of pancreatitis who no longer require treatment for diabetes are eligible.
* Known osteoporosis or receipt of treatment of osteopenia or osteoporosis within 12 weeks prior to study entry with the following medications: risedronate (Actonel®), ibandronate (Boniva®), etidronate (Didronel®), raloxifene (Evista®), teriparatide (Forteo®), aledronate (Fosamax®), calcitonin (Miacalcin®).
* Inability to tolerate consumption of an ice cream-based milkshake.
* Regular and excessive use of alcohol defined as self-reported alcohol intake >120 g of alcohol/week in a male or >60 g alcohol/week in a female within 12 weeks immediately prior to study entry.
* Unwilling to restrict alcohol use during the study to ≤120g alcohol/week in a male or ≤60 g alcohol/week in a female.
* Unwilling to restrict diet during the study (both Step 1 and Step 2).
* Known glucocorticoid use in supraphysiologic doses (prednisone >10 mg/day or equivalent doses of other glucocorticoids) within 12 weeks prior to study entry.
* Known glucocorticoid use in physiologic replacement doses (prednisone ≤10 mg/day or equivalent doses of other glucocorticoids) initiated within 28 days prior to study entry. NOTE: Individuals on physiologic replacement doses of glucocorticoids initiated more than 28 days prior to study entry will not be excluded.
* History of congestive heart failure corresponding to New York Heart Association Class II or greater
* Current use of prohibited concomitant medications
* Current participation in experimental studies that include treatments not approved by the FDA or any blinded treatments.
* Body mass index (BMI) > 35 kg/m2.
* Known allergy to food contained within the standard meal (i.e. chicken, soy)
* Subjects with a history of clinically significant cardiac disease, including a family history of Long QT Syndrome, and/or evidence of the following ECG abnormalities at screening:

  * QTcF (QT corrected using Fridericia's formula, Fridericia's formula: QTcF=QT/(RR^0.333) of > 450 msec; complete or incomplete left or right bundle branch block; intraventricular conduction delay with QRS duration of > 120 msec; bradycardia (< 45 beats per minute);
  * pathologic Q-waves (Q-wave of > 40 msec or depth of > 0.4 to 0.5 V);
  * arrhythmia (an isolated premature ventricular contraction on screening/Day 1 is not exclusionary) ;
  * ventricular pre-excitation;
  * second or third degree heart block.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Naringenin pharmacokinetic curves | 12 hours
  Level of naringenin will be measured by HPLC at time 0, 30, 40, 90, 120, 150, and 180 min and at 4, 5, 6, 7, 8, and 12 hours.

SECONDARY OUTCOMES:
Safety | 12 hours
  as indicated by all high-grade signs and symptoms and laboratory values.
Changes in HCV RNA levels | 12 hours
Homeostatic model assessment-insulin resistance (HOMA-IR) | 24 hours
Lipid levels: Cholesterol and triglyceride levels | 24 hours
Liver enzyme levels | 24 hours
  ALT and AST at entry and end of steps 1 and 2.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Y Kim, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Nahmias Y, Goldwasser J, Casali M, van Poll D, Wakita T, Chung RT, Yarmush ML. Apolipoprotein B-dependent hepatitis C virus secretion is inhibited by the grapefruit flavonoid naringenin. Hepatology. 2008 May;47(5):1437-45. doi: 10.1002/hep.22197. PMID 18393287